CLINICAL TRIAL: NCT04461808
Title: Tomosynthesis as Primary Test for Breast Cancer Screening: A Multicenter Randomized Controlled Trial
Brief Title: Tomosynthesis as Primary Test for Breast Cancer Screening
Acronym: MAITA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Collaborators: AULSS 9 Scaligera di Verona (Unknown); IRCCS Policlinico S. Donato, Milano (Unknown); Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: RF-2016-02363686
Record Dates: First submitted 2020-07-01; First posted 2020-07-08 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: breast cancer screening; tomosynthesis
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Intervention Model Description: Women 45-65 participating in the mammographic screening program will be randomized to one round of screening with tomosynthesis + synthetic 2D or with digital mammography. Then all women will be re-screened after 2 years (1 year for women 45-49) for at least one round with digital mammography.
Who Masked: Outcomes Assessor
Masking Description: It is not possible to mask the intervention for the patient, care provider, and investigator.
  Only the assessment of one of the two co-primary outcomes, i.e. cumulative incidence of advanced breast cancer after the first round of screening, can be masked. This will be obtained through a blind review of an external panel of pathologists and radiologists reviewing cases retrieved by cancer registries.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tomosynthesis + synthetic 2D (Experimental): Women will be screened for one round with tomosynthesis + synthetic 2D, two projections, double reading with consensus or arbitration, according to local protocols, for discordant readings.
  After two years (one years for women 45-49 yo) women will be re-screened with digital mammography.
  Interventions: Diagnostic Test: tomosynthesis + synthetic 2D
- Digital Mammography (Active Comparator): Women will be screened for digital mammography, two projections, double reading with consensus or arbitration, according to local protocols, for discordant readings.
  After two years (one years for women 45-49 yo) women will be re-screened with digital mammography.
  Interventions: Diagnostic Test: digital mammography

INTERVENTIONS:
Diagnostic Test: tomosynthesis + synthetic 2D — Women will be screened for one round with tomosynthesis + synthetic 2D, two projections, double reading with consensus or arbitration, according to local protocols, for discordant readings.
  After two years (one years for women 45-49 yo) women will be re-screened with digital mammography.
  Arms: Tomosynthesis + synthetic 2D
Diagnostic Test: digital mammography — Women will be screened for one round digital mammography, two projections, double reading with consensus or arbitration, according to local protocols, for discordant readings.
  After two years (one years for women 45-49 yo) women will be re-screened with digital mammography.
  Arms: Digital Mammography

SUMMARY:
Randomized trial comparing tomosynthesis plus synthetic 2D Mammography vs Digital Mammography in respect to incidence of advanced cancers (interval and following round) and interval cancers.

DETAILED DESCRIPTION:
This is a companion study of the other Italian studies on tomosyntesis as primary screening test for breast cancer: RETomo (NCT02698202), PROTEUS (NCT02590315), IMPETO (NCT03587259). The investigators conduct a randomized trial in three centres with a protocol that is similar to that of the other three studies. As for IMPETO and differently from the RETomo and PROTEUS studies, the intervention will be tomosynthesis + synthetic 2D.

In the three centres about 8000 women will be recruited (4000 in the experimental arm and 4000 in the control arm).

The study will compare the performance of tomosynthesis plus synthetic 2D vs digital mammography in respect to incidence of advanced cancers (interval and following round) and interval cancers. Women 50 to 65 years old will be screened once according to randomization arm for one round, then all will be screened with digital mammography after two years.

The investigators also will measure detection rates, specificity, interval cancers, advanced cancers occurring as interval cancers or at subsequent screens and allowing to estimate excess overdiagnosis comparing overall cumulative incidence after two or three rounds of screening.

Women will be asked for informed consent when they attend the mammography. If they accept they will be randomised to one of the two arms.

All examinations will be read by two independent radiologists, in case of discordance a third reading is asked.

ELIGIBILITY:
Inclusion Criteria:

* Women scheduled for a new round of mammographic screening
* resident in the province

Exclusion Criteria:

* previous breast cancer diagnosis
* pregnancy or suspicion of pregnancy
* presence of BRCA1/2 gene mutation
* Previous Digital Breast Tomosynthesis performed
* unable to understand informed consent
* chemotherapy in progress
* presence of breast implant

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10156 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
advanced cancer incidence | 2 years (+9 months to complete second round assessment)
  cumulative incidence of T2+ cancers after first screening round
advanced cancer incidence | 4 years (+9 months to complete third round assessment)
  cumulative incidence of T2+ cancers after first screening round
interval cancer incidence | 2 years for 50-65 years old women
  incidence of cancers occurring after a negative screening test and before the next scheduled screening round. Outcome 3 and 4 will are combined in one single outcome.
interval cancer incidence | 1 year for 45-49 years old women
  incidence of cancers occurring after a negative screening test and before the next scheduled screening round. Outcome 3 and 4 will are combined in one single outcome.

SECONDARY OUTCOMES:
overall cumulative incidence | 2 years (+9 months to complete second round assessment)
  overall cumulative incidence of breast cancer, including ductal carcinoma in situ. This outcome is a proxy of the excess over-diagnosis eventually induced by tomosynthesis compared with digital mammography.
overall cumulative incidence | 4 years (+9 months to complete second round assessment)
  overall cumulative incidence of breast cancer, including ductal carcinoma in situ. This outcome is a proxy of the excess over-diagnosis eventually induced by tomosynthesis compared with digital mammography.
detection rate | This outcome is measured at the baseline screening. cancer diagnosed within 9 months will be considered
  cancer detected by the screening round on total screened women
recall rate | This outcome is measured at the baseline screening.
  number of women referred to assessment after the first leve screening test on total screened women
positive predictive value | This outcome is measured at the baseline screening. cancer diagnosed within 9 months will be considered
  proportion of cancer among women recalled for assessment
Detection rate of ductal carcinoma in situ | This outcome is measured at the baseline screening. cancer diagnosed within 9 months will be considered
  ductal carcinoma in situ detected by the screening round on total screened women
biopsy rate | This outcome is measured at the baseline screening.
  number of women undergoing biopsy after the first leve screening test on total screened women
x-ray dose | This outcome is measured at the baseline screening.
  average glandular dose receive by women during first level test
reading time | This outcome is measured at the baseline screening.
  time needed to read an imaging first level examination

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Azienda Unità Sanitaria Locale - IRCCS di Reggio Emilia, Reggio Emilia, Italy
  - IRCCS Policlinico San Donato, Milan
  - Azienda Ospedaliera Universitaria Integrata, Verona
  - Azienda Ulss 9 Scaligera, Verona